CLINICAL TRIAL: NCT07063784
Title: Patient Positioning for Hand, Wrist, and Elbow Surgery: Stretcher Versus Operating Room Table, A Randomized Controlled Trial
Brief Title: Patient Positioning for Hand, Wrist, and Elbow Surgery: Stretcher Versus Operating Room Table
Status: Completed | Type: Observational
Sponsor: Brett Lewellyn (Other)
Responsible Party: Sponsor-Investigator, Brett Lewellyn, Chief Hand & Upper Extremity Surgery, Orlando Health, Inc.
Organization: Orlando Health, Inc. (Other)
Other Study IDs: 17.048.05
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Post-operative Complications; Operative Surfaces

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients randomized to undergo surgery on an OR table
- patients randomized to undergo surgery on a stretcher with a hand table

SUMMARY:
The purpose of this study is to determine if there is any difference with regard to complication rates for performing surgery on an operating room (OR) table vs performing surgery on a stretcher with a hand table. The OR table and the stretcher with a hand table are the two types of operative surfaces the investigators will compare. The aim of this study is to compare surgeries of finger, hand, wrist, forearm, and elbow. The investigators will conduct the research at two outpatient surgery centers and an inpatient hospital center to see if operating room surface and time of surgery has any effect on complications after surgery. The investigators also will compare the costs of the two types of operative surfaces for the surgery.

DETAILED DESCRIPTION:
The primary objective is to determine if there is any difference with regard to complication rate for performing surgery on an OR table vs performing surgery on a stretcher with a hand table. Outcome measures will include any complications recorded by postoperative questionnaires filled out by patients, and examination of the data to see if there is any statistically significant (using P values) data.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will involve skeletally mature adult patients who are to be operated on by the principal investigator, in a one year time frame, for any surgical procedure of the upper extremity from the fingertip to the middle portion of the arm above the elbow.

Exclusion Criteria:

* Exclusion criteria will include: the skeletally immature, any patient with pre-existing neck pain, back pain, or decubitus ulcers; and patients with preexisting "pain" related or other conflicting medical issues: i.e. fibromyalgia; patients who were unable to respond for themselves in postop follow up i.e. dementia, Parkinson's disease, Alzheimer's and stroke.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: two outpatient surgery centers and an inpatient hospital center
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine if there are increased or decreased complications when comparing patients who are having surgical procedures on an OR table vs a standard hospital stretcher. | From enrollment to one year postoperative

SECONDARY OUTCOMES:
This will include determining any correlation between surgical time, length of follow up and complication rate according to surgical procedure and operating surface. | From enrollment to one year postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No